CLINICAL TRIAL: NCT02709850
Title: A Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of ISIS 703802, Targeting ANGPTL3, Administered Subcutaneously to Healthy Volunteers With Elevated Triglycerides and Subjects With Familial Hypercholesterolemia
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IONIS ANGPTL3-LRx in Healthy Volunteers With Elevated Triglycerides and Participants With Familial Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ISIS 703802-CS1; 2015-004003-23 (EudraCT Number)
Record Dates: First submitted 2015-11-22; First posted 2016-03-16 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Hypertriglyceridemia; Familial Hypercholesterolemia
Keywords: ANGPTL-3
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type II | interventions — IONIS-ANGPTL3-LRx

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohorts A, D: Placebo (Placebo Comparator): Participants received a single-dose of IONIS ANGPTL3-LRx-matching placebo subcutaneously on Day 1.
  Interventions: Drug: Placebo
- Cohorts A, D: IONIS ANGPTL3-LRx 20 mg (Experimental): Participants received a single-dose of IONIS ANGPTL3-LRx 20 milligrams (mg) subcutaneously on Day 1.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts A, D: IONIS ANGPTL3-LRx 120 mg (Experimental): Participants received a single-dose of IONIS ANGPTL3-LRx 120 mg subcutaneously on Day 1.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts B, C: Placebo (Placebo Comparator): Participants received a single-dose of IONIS ANGPTL3-LRx-matching placebo subcutaneously on Day 1.
  Interventions: Drug: Placebo
- Cohorts B, C: IONIS ANGPTL3-LRx 40 mg (Experimental): Participants received a single-dose of IONIS ANGPTL3-LRx 40 mg subcutaneously on Day 1.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts B, C: IONIS ANGPTL3-LRx 80 mg (Experimental): Participants received a single-dose of IONIS ANGPTL3-LRx 80 mg subcutaneously on Day 1.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts AA-DD: Placebo (Placebo Comparator): Participants received IONIS ANGPTL3-LRx-matching placebo subcutaneously once per week for 6 weeks.
  Interventions: Drug: Placebo
- Cohorts AA-DD: IONIS ANGPTL3-LRx 10 mg (Experimental): Participants received IONIS ANGPTL3-LRx 10 mg subcutaneously once per week for 6 weeks.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts AA-DD: IONIS ANGPTL3-LRx 20 mg (Experimental): Participants received IONIS ANGPTL3-LRx 20 mg subcutaneously once per week for 6 weeks.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts AA-DD: IONIS ANGPTL3-LRx 40 mg (Experimental): Participants received IONIS ANGPTL3-LRx 40 mg subcutaneously once per week for 6 weeks.
  Interventions: Drug: IONIS ANGPTL3-LRx
- Cohorts AA-DD: IONIS ANGPTL3-LRx 60 mg (Experimental): Participants received IONIS ANGPTL3-LRx 60 mg subcutaneously once per week for 6 weeks.
  Interventions: Drug: IONIS ANGPTL3-LRx

INTERVENTIONS:
Drug: IONIS ANGPTL3-LRx
  Other Names: ISIS 703802
  Arms: Cohorts A, D: IONIS ANGPTL3-LRx 120 mg; Cohorts A, D: IONIS ANGPTL3-LRx 20 mg; Cohorts AA-DD: IONIS ANGPTL3-LRx 10 mg; Cohorts AA-DD: IONIS ANGPTL3-LRx 20 mg; Cohorts AA-DD: IONIS ANGPTL3-LRx 40 mg; Cohorts AA-DD: IONIS ANGPTL3-LRx 60 mg; Cohorts B, C: IONIS ANGPTL3-LRx 40 mg; Cohorts B, C: IONIS ANGPTL3-LRx 80 mg
Drug: Placebo — 0.9%NaCl, water, riboflavin
  Arms: Cohorts A, D: Placebo; Cohorts AA-DD: Placebo; Cohorts B, C: Placebo

SUMMARY:
The purpose is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of IONIS ANGPTL3-LRx (ISIS 703802) given to healthy volunteer subjects with elevated triglycerides and subjects with familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria for All Cohorts:

* Must have given written informed consent and be able to comply with all study requirements
* Males or females 18 to 65 years, inclusive, at the time of informed consent
* Body Mass Index (BMI) ≤ 35.0 kg/m2
* Females must be non-pregnant and non-lactating, and either surgically sterile or postmenopausal.
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method

Inclusion criteria for Cohorts, A, D, and AA to DD only:

* Fasting triglycerides (TG) ≥ 150 mg/dL at Screening
* Fasting low density lipoprotein cholesterol (LDL-C) > 70 mg/dL at Screening

Inclusion criteria for Cohorts B and C only:

* Fasting TG 90 - 150 mg/dL at Screening
* Fasting LDL-C > 70 mg/dL at Screening

Inclusion Criteria for Cohort EE Only:

* Homozygous FH diagnosis and fasting LDL-C ≥ 190 mg/dL (4.9 mmol/L)

Inclusion Criteria for Cohort FF Only:

* Heterozygous FH diagnosis and fasting LDL-C ≥ 160 mg/dL (4.1 mmol/L)

Inclusion Criteria for Cohorts EE and FF Only:

* Maximally tolerated stable LDL-C lowering agents (stable for at least 12 weeks)
* On stable low-fat diet
* Stable weight (± 4 kg) for ≥ 6 weeks prior to screening

Exclusion Criteria for All Cohorts:

* Known history or positive test for Human Immunodeficiency Virus (HIV), Hepatitis C (HCV), or Hepatitis B (HBV)
* Treatment with another Study Drug, biological agent, or device within one-month or 5-half-lives of screening
* Regular use of alcohol within 6 months of screening
* Use of concomitant drugs unless authorized by the Sponsor Medical Monitor
* Known contraindication and/or allergy to heparin
* Smoking > 10 cigarettes a day
* Considered unsuitable for inclusion by the Principal Investigator

Exclusion Criteria for Cohorts EE and FF:

* Myocardial infarction, percutaneous transluminal coronary intervention, or coronary artery bypass graft surgery within 12 weeks prior to screening, or cerebrovascular accident within 24 weeks prior to screening. Participants with adequately treated stable angina, per Investigator assessment, may be included
* Congestive heart failure defined by NYHA Classes III or IV
* Type 2 diabetes mellitus (T2DM) with HbA1c > 8.0%
* Prior treatment with gene therapy
* Currently receiving apheresis treatments or last apheresis treatment was within 8 weeks of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of IONIS ANGPTL3-LRx (incidence, severity, and dose-relationship of adverse effects and changes in the laboratory parameters) | Up to Day 127
  The safety and tolerability of IONIS ANGPTL3-LRx will be assessed by determining the incidence, severity, and dose-relationship of adverse effects and changes in the laboratory parameters by dose. Safety results in subjects dosed with IONIS ANGPTL3-LRx will be compared with those from subjects dosed with placebo.
Pharmacokinetics after single and multiple doses of IONIS ANGPTL3-LRx. | Up to Day 127
  The plasma pharmacokinetics (concentration-time results) of IONIS ANGPTL3-LRx (unconjugated and conjugated ASO) will be assessed following single and multiple-dose SC administration. The amount of IONIS ANGPTL3-LRx excreted in urine at selected 24-hour intervals will also be determined.
Pharmacodynamics of IONIS ANGPTL3-LRx (Changes in serum ANGPTL3 levels) | Up to Day 127
  Changes in serum angiopoietin-like 3 (ANGPTL3) levels compared to baseline.

SECONDARY OUTCOMES:
Pharmacodynamic effects of IONIS ANGPTL3-LRx | Up to Day 127
  Effects of IONIS ANGPTL3-LRx on changes in ANGPTL3 plasma protein compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graham MJ, Lee RG, Brandt TA, Tai LJ, Fu W, Peralta R, Yu R, Hurh E, Paz E, McEvoy BW, Baker BF, Pham NC, Digenio A, Hughes SG, Geary RS, Witztum JL, Crooke RM, Tsimikas S. Cardiovascular and Metabolic Effects of ANGPTL3 Antisense Oligonucleotides. N Engl J Med. 2017 Jul 20;377(3):222-232. doi: 10.1056/NEJMoa1701329. Epub 2017 May 24. PMID 28538111